CLINICAL TRIAL: NCT01359917
Title: Psychological Morbidity and Facial Volume in HIV Lipodystrophy:
Brief Title: Psychological Morbidity and Facial Volume in HIV Lipodystrophy: Quantification of Treatment Outcome
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Dr Lisa Nelson, NHS Lothian
Other Study IDs: REC06/MRE00/39
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2006-03

CONDITIONS: HIV-Associated Lipodystrophy Syndrome
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- autologous fat transfer: patients received fat transfer for HIV lipodystrophy
- polylactic acid: treatment with polylactic acid (PLA) for HIV lipodystrophy
- bio-alcamid: bio-alcamid injections

SUMMARY:
The hypotheses of this study were that:

1. HIV lipodystrophy is associated with psychological morbidity relating to body image, anxiety and depression.
2. Treatment of HIV lipodystrophy using autologous fat transfer, polylactic acid or Bio-alcamid, is associated with an improvement in psychological morbidity and anatomical volume of treated areas.
3. The DI3D system is a valid and reproducible method of recording and measuring facial 3-D volume.

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

* HIV facial lipoatrophy
* concurrent antiretrovirals

Exclusion Criteria:

* known psychological disorder
* skin allergies
* significant medical problems precluding anaesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with HIV facial lipoatrophy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
measurement of 3-D facial volume | 2 years
  3-D facial camera

SECONDARY OUTCOMES:
psychological outcome | 2 years
  derriford appearance scale hospital anxiety and depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Stewart, FRCSPlast, Principal Investigator — NHS Lothian

REFERENCES:
- [Derived] Nelson L, Stewart KJ. Psychological morbidity and facial volume in HIV lipodystrophy: quantification of treatment outcome. J Plast Reconstr Aesthet Surg. 2012 Apr;65(4):439-47. doi: 10.1016/j.bjps.2011.11.024. Epub 2011 Dec 5. PMID 22153841